CLINICAL TRIAL: NCT01049334
Title: A Randomized, Double-Blind, Placebo-Controlled Multiple-Dose Study to Determine the Efficacy, Onset, and Duration of Action of Flurbiprofen 8.75 mg Lozenge Compared to Its Vehicle Control Lozenge in Patients With Painful Pharyngitis
Brief Title: A Study of Flurbiprofen 8.75 mg Lozenge in Patient With Pharyngitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Reckitt Benckiser LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TH 0901
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Results first posted 2017-09-21 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-08

CONDITIONS: Pharyngitis
MeSH Terms: conditions — Pharyngitis | interventions — Flurbiprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- flurbiprofen 8.75 mg lozenge (Experimental): Participants sucked flurbiprofen 8.75mg lozenge every 3-6 hours up to 5 lozenges a day as needed for pain for 7 days.
  Interventions: Drug: Flurbiprofen
- Placebo lozenge (Placebo Comparator): Participants sucked vehicle placebo lozenge every 3-6 hours up to 5 lozenges a day as needed for pain for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Participants were instructed to suck one placebo lozenge during the initial two-hour clinic visit. Upon discharge, participants were instructed to use study medication lozenge every 3-6 hours as needed for pain, up to a total of 5 study lozenges in 24 hours.
  Arms: Placebo lozenge
Drug: Flurbiprofen — Participants were instructed to suck one flurbiprofen 8.75 mg lozenge during the initial two-hour clinic visit. Upon discharge, participants were instructed to use study medication lozenge every 3-6 hours as needed for pain, up to a total of 5 study lozenges in 24 hours.
  Arms: flurbiprofen 8.75 mg lozenge

SUMMARY:
The purposes of this study is to demonstrate the analgesic efficacy of flurbiprofen 8.75 mg lozenge compared to its vehicle lozenge and to demonstrate the safety of the flurbiprofen lozenge throughout the course of treating sore throat due to acute pharyngitis.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a complaint of sore throat.
2. If the patient is a female of childbearing potential, she has been using effective contraception since the last date of menses and is not breast-feeding or lactating.
3. If the patient is a female of childbearing potential, the patient must have a negative urine pregnancy.
4. The patient has provided written informed consent prior to any study-related procedures.

Exclusion Criteria:

1. The patient has a history of an upper gastrointestinal ulcer within the past 60 days, is currently experiencing clinically significant upper gastrointestinal complaints, or is currently taking medication regularly (≥ three times in the previous week).
2. The patient has a history of any hepatic disease or renal dysfunction.
3. The patient has a history of chronic analgesic use (≥ three times per week over the prior four weeks). (Patients on low-dose aspirin therapy may be allowed in the study per investigator's clinical decision.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Shea, BS, Study Director — Reckitt Benckiser Inc.
Locations (1):
- University of Connecticut, Student Health Services, Storrs, Connecticut, United States

REFERENCES:
- [Result] Schachtel BP, McCormick CG and Giefer EE. Patient-reported outcomes (PRO's) in the pharyngitis pain model. Abstract presented at the International Association for the Study of Pain (IASP) Scientific Conference, Montreal, Canada. 2009
- [Result] Schachtel BP, Aspley S, Sternberg M, Berry P, Muir N, Sanner K, Rezuke J, Savino L, Shephard A, Shea T, Schachtel E. Onset of demulcent and analgesic activity of flurbiprofen lozenge. Int J Clin Pharm 2012;34:143-258.
- [Result] Aspley S, Schachtel B, Berry P, Shephard A, Sanner K, Shea T, Smith G. The Chief Complaint: evidence of its use as an endpoint in a clinical trial. Journal of Pain 2012;13(4)Supplement:S4.
- [Result] Aspley S, Schachtel B, Berry P, Shephard A, Sanner K, Savino L, Rezuke J, Shea T, Smith G. Treatment of odynophagia and dysphagia by flurbiprofen 8.75 mg lozenges. Pain Research & Management 2012;17(3):203.
- [Result] Schachtel B, Aspley S, Berry P, Shephard A, Shea T,Sanner K, Smith G,Schachtel E. Efficacy of flurbiprofen 8.75mg lozenges in patients with swollen/inflamed sore throat. Abstract presented at the 14th World Congress on Pain, 27 - 31 August 2012, Milan.
- [Result] Schachtel B, Aspley S, Berry P, Smith G, Shephard A, Shea T, Schachtel E. A patient-centered method for determining onset of action. Clinical Pharmacology in Drug Development 2012;1(4):194-195.
- [Result] Schachtel B, Aspley S, Berry P, Shephard A, Shea T, Smith G, Sanner K, Savino L, Rezuke J, Schachtel E. Efficacy and duration of flurbiprofen 8.75 mg lozenge. Clinical Pharmacology in Drug Development 2012;1(4):194.
- [Result] Schachtel B, Aspley S, Berry P, Shephard A, Shea T, Smith G, Schachtel E. A new cough model: de-hawthornizing a clinical trial. Clinical Pharmacology in Drug Development 2012;1(4):195.
- [Result] Schachtel B, Aspley S, Berry P, Shephard A, Sanner K, Shea T, Smith G, Schachtel E. Chief Complaint: the therapeutogenic stimulus as the primary, individualized endpoint in clinical trials. Journal of Pain 2012;13(4)Supplement:S6.
- [Result] Aspley S, Schachtel B, Berry P, Shephard A, Shea T, Smith G, Schachtel E. Flurbiprofen lozenges in patients with a "bad sore throat". Journal of Pain 2013;14(4):S59.
- [Result] Schachtel B, Aspley S, Berry P, Shephard A, Shea T, Smith G, Schachtel E. The "Definite Improvement Level" (DIL) as a determinant of drug efficacy. Journal of Pain 2013;14(4):S5.
- [Result] Shephard A, Smith G, Aspley S, Schachtel B. Efficacy of flurbiprofen 8.75 mg lozenges for streptococcal and non-streptococcal sore throat: pooled analysis of two randomised, placebo-controlled studies. Abstract presented at the European Congress of Clinical Microbiology and Infectious Diseases (ECCMID), 27 - 30 April 2013, Berlin.
- [Result] Shephard A, Smith G, Aspley S, Schachtel B. Symptomatic relief in streptococcal and non-streptococcal sore throat patients: pooled analysis of two randomised, placebo-controlled studies. Abstract presented at the European Congress of Clinical Microbiology and Infectious Diseases (ECCMID), 27-30 April 2013, Berlin.
- [Derived] Aspley S, Shephard A, Schachtel E, Sanner K, Savino L, Schachtel B. Efficacy of flurbiprofen 8.75 mg lozenge in patients with a swollen and inflamed sore throat. Curr Med Res Opin. 2016 Sep;32(9):1529-38. doi: 10.1080/03007995.2016.1187119. Epub 2016 May 18. PMID 27146963
- [Derived] Shephard A, Smith G, Aspley S, Schachtel BP. Randomised, double-blind, placebo-controlled studies on flurbiprofen 8.75 mg lozenges in patients with/without group A or C streptococcal throat infection, with an assessment of clinicians' prediction of 'strep throat'. Int J Clin Pract. 2015 Jan;69(1):59-71. doi: 10.1111/ijcp.12536. Epub 2014 Oct 9. PMID 25296661

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two hundred twenty-seven patients were screened.
Period: Overall Study
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Started | 102 | 102
Completed | 93 | 95
Not Completed | 9 | 7
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Adverse Event | 2 | 3
Not completed — Physician Decision | 2 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge | Total
Number analyzed (Participants) | 102 | 102 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.8 (1.48) | 19.8 (1.47) | 19.8 (1.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 63 | 117
  Male | 48 | 39 | 87
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 96 | 97 | 193
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African | 5 | 2 | 7
  White | 92 | 95 | 187
  Multi-racial | 0 | 1 | 1
  Other, not specified | 2 | 2 | 4
Sore Throat Pain Intensity Scale (STPIS) [Mean (Standard Deviation); unit: units on a scale] — STPIS measures sore throat pain intensity on a 100-mm visual analog scale completed by participants. A mark at 0-mm indicates no pain upon swallowing and 100-mm indicates severe pain.
  units on a scale | 78.8 (8.56) | 80.5 (7.92) | 79.7 (8.27)
Difficulty Swallowing Scale (DSS) [Mean (Standard Deviation); unit: units on a scale] — Participants were asked to evaluate his/her difficulty swallowing (dysphagia) using a 100-mm visual analog scale. Participants were instructed to swallow and "Place a line on the scale that best characterizes how difficult it is to swallow now." A mark at 0-mm indicated no difficulty and 100-mm indicated very difficult.
  units on a scale | 76.9 (12.41) | 76.3 (11.04) | 76.6 (11.72)
Swollen Throat Scale (SwoTS) [Mean (Standard Deviation); unit: units on a scale] — he participant was asked to evaluate how swollen his/her throat felt using a 100-mm visual analog scale. The patient was instructed to swallow and "Place a line on the scale that best characterizes how swollen your throat feels now." A mark at 0-mm indicated not swollen and 100-mm indicated very swollen.
  units on a scale | 76.6 (13.98) | 79.0 (12.05) | 77.8 (13.07)

OUTCOME MEASURES:

1. Primary Outcome: Time Weighted Sum of Pain Intensity Differences (SPID) in Sore Throat Pain Intensity Scale (STPIS) Over the 24 Hours Post-baseline (STPIS SPID24)
Description: STPIS measures sore throat pain intensity on a 100-mm visual analog scale completed by participants. A mark at 0-mm indicates no pain upon swallowing and 100-mm indicates severe pain. SPID24 was calculated as the sum of the time-weighted pain intensity differences from baseline until 24 hours. The full range was -114609 (complete pain relief within 2 minutes of dosing that lasts 24 hours) to 29191 (maximum pain within 2 minutes lasting 24 hours) using the mean baseline STPIS. Participants with a last recorded time point <21 hours were considered Not Evaluable. If a participant used rescue medication, all post-rescue STPIS values in the 24-hour interval were assigned the baseline value for STPIS. Missing scores of STPIS with non-missing STPIS scores at earlier and later assessments were imputed using linear interpolation assuming the time of the missing assessment to be the nominal time since initial dose.
Time Frame: baseline (pre-dose), 24 hours post-dose (every 2 minutes for one hour; every 10 minutes until hour 2; every 30 minutes until hour 6; and every hour the participant was awake between hours 7-24)
Population: Intent to treat population of participants who took the first full dose of medication. Three participants (1 Flurbiprofen, 2 Placebo) did not have sufficient 24 hour data to be included in the primary analysis of the primary endpoint (no entries after 2 hours), but did have sufficient data to be included in other efficacy analyses.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 101 | 100
units on a scale | -473.7 (45.4428) | -322.3 (45.6708)
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.0201, ANOVA — The a priori threshold for statistical significance is 0.05. No adjustments for statistical multiplicity were required; Treatment as a fixed effect and baseline STPIS as a covariate; least-square means difference = -151.5, 95% CI 2-sided [-278.9 to -24.0]

2. Secondary Outcome: Time Weighted Sum of Pain Intensity Differences (SPID) in Sore Throat Pain Intensity Scale (STPIS) Over the 2 Hours Post-baseline (STPIS SPID2)
Description: STPIS measures sore throat pain intensity on a 100-mm visual analog scale completed by participants. A mark at 0-mm indicates no pain upon swallowing and 100-mm indicates severe pain. SPID2 was calculated as the sum of the time-weighted pain intensity differences from baseline until 2 hours post dosing. The full range was -9405 (complete pain relief within 2 minutes of dosing that lasts 2 hours) to 2395 (maximum pain within 2 minutes lasting 2 hours) using the mean baseline STPIS.
  If a participant used rescue medication (acetaminophen 650mg was allowed as needed post dose), all post-rescue STPIS values in the 24-hour interval were assigned the baseline value for STPIS. Missing scores of STPIS with non-missing STPIS scores at earlier and later assessments (recorded or derived due to rescue) were imputed using linear interpolation assuming the time of the missing assessment to be the nominal time since initial dose.
Time Frame: baseline (pre-dose), 2 hours post-dose (every 2 minutes for one hour; every 10 minutes until hour 2)
Population: Intent to treat population of participants who took the first full dose of medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 102 | 102
units on a scale | -43.4 (39.20) | -23.5 (29.52)
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p < .0001, ANOVA — The a priori threshold for statistical significance is 0.05. Closed-sequential approach to control type I error: analyses through secondary outcomes #2-13 in the order listed will proceed until a p-value >0.05 occurs; Treatment as a fixed effect and baseline of the variable predicted as a covariate; least-square means difference = -19.6, 95% CI 2-sided [-29.2 to -9.9]

3. Secondary Outcome: Time Weighted Summed Differences in Difficulty Swallowing Scale (DSS) During the Initial 2 Hours From Baseline
Description: Participants were asked to evaluate his/her difficulty swallowing (dysphagia) using a 100-mm visual analog scale at Baseline and 2 hours post dose.
  Participants were instructed to swallow and "Place a line on the scale that best characterizes how difficult it is to swallow now." A mark at 0-mm indicated no difficulty and 100-mm indicated very difficult. Data is reported as the sum of the time-weighted pain intensity differences from baseline until 2 hours post dose. The full range was -9192 (no difficulty swallowing within 10 minutes of dosing that lasts 2 hours) to 2808 (maximum difficulty swallowing within 10 minutes lasting 2 hours) using the baseline DSS value.
  Missing values of DSS with non-missing values at assessments before and after were calculated using linear interpolation.
Time Frame: baseline (pre-dose), 2 hours post-dose (every 10 minutes until hour 2)
Population: Intent to treat population of participants who took the first full dose of medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 102 | 102
units on a scale | -39.1 (38.64) | -16.6 (29.34)
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 2, analysis 1]; Treatment as a fixed effect and baseline of the variable predicted as a covariate; least-square means difference = -22.3, 95% CI 2-sided [-31.7 to -12.9]

4. Secondary Outcome: Time Weighted Summed Differences in Difficulty Swallowing Scale (DSS) During the Initial 24 Hours From Baseline
Description: Participants were asked to evaluate his/her difficulty swallowing (dysphagia) using a 100-mm visual analog scale at Baseline and until 24 hours post dose.
  Participants were instructed to swallow and "Place a line on the scale that best characterizes how difficult it is to swallow now." A mark at 0-mm indicated no difficulty and 100-mm indicated very difficult. Data is reported as the sum of the time-weighted pain intensity differences from baseline until 24 hours post dose. The full range was -110304 (no difficulty swallowing within 10 minutes of dosing that lasts 24 hours) to 33696 (maximum difficulty swallowing within 10 minutes lasting 24 hours) using the baseline DSS value.
  Missing values of DSS with non-missing values at assessments before and after were calculated using linear interpolation.
Time Frame: baseline (pre-dose), 24 hours post-dose (every 10 minutes until hour 2, every 30 minutes until hour 6, hourly from 7-24 hours)
Population: Intent to treat population of participants who took the first full dose of medication and had DSS recorded after 21-hours.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 101 | 99
units on a scale | -460.8 (498.79) | -274.3 (455.35)
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.0071, ANOVA — [p-value comment as in outcome 2, analysis 1]; Treatment as a fixed effect and baseline of the variable predicted as a covariate; least-square means difference = -181.7, 95% CI 2-sided [-313.7 to -50.0]

5. Secondary Outcome: Time Weighted Summed Differences in Swollen Throat Scale (SwoTS) During the Initial 2 Hours From Baseline
Description: The participant was asked to evaluate how swollen his/her throat felt using a 100-mm visual analog scale at Baseline and at 1 hour, 70 minutes, 80 minutes, 90 minutes, 100 minutes, 110 minutes, and 2 hours.
  The patient was instructed to swallow and "Place a line on the scale that best characterizes how swollen your throat feels now." A mark at 0-mm indicated not swollen and 100-mm indicated very swollen. The full range of the sum of the time-weighted swollen throat differences from baseline until 2 hours was -9336 (throat did not feel swollen at all within 1 hour of dosing and lasted 2 hours) to 2664 (maximum swollen throat reported within 1 hour and lasting 2 hours) using the mean baseline SwoTS.
Time Frame: baseline (pre-dose), 2 hours post-dose (at 1 hour, 70 minutes, 80 minutes, 90 minutes, 100 minutes, 110 minutes, and 2 hours)
Population: Intent to treat population of participants who took the first full dose of medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 102 | 102
units on a scale | -39.9 (39.63) | -20.1 (27.28)
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 2, analysis 1]; Treatment as a fixed effect and baseline of the variable predicted as a covariate; least-square means difference = -20.8, 95% CI 2-sided [-30.2 to -11.2]

6. Secondary Outcome: Time Weighted Summed Differences in Swollen Throat Scale (SwoTS) During the Initial 24 Hours From Baseline
Description: The participant was asked to evaluate how swollen his/her throat felt using a 100-mm visual analog scale at Baseline and specified timeframes until 24 hours.
  The patient was instructed to swallow and "Place a line on the scale that best characterizes how swollen your throat feels now." A mark at 0-mm indicated not swollen and 100-mm indicated very swollen. The full range of the sum of the time-weighted swollen throat differences from baseline until 24 hours was -112032 (throat did not feel swollen at all within 1 hour of dosing and lasted 24 hours) to 31968 (maximum swollen throat reported within 1 hour and lasting 24 hours) using the mean baseline SwoTS.
Time Frame: baseline (pre-dose), 24 hours post-dose (1 hour, 70 minutes, 80 minutes, 90 minutes, 100 minutes, 110 minutes, 2 hours, 2½ hours, 3 hours, 3½ hours, 4 hours, 4½ hours, 5 hours, 5½ hours, and 6 hours after the first dose, hourly from 7-24 hours)
Population: Intent to treat population of participants who took the first full dose of medication, and had SwoTS recorded after 21 hours. Four participants (1 Flurbiprofen, 3 Vehicle) did not have SwoTS recorded after 21 hours and were not included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 101 | 99
units on a scale | -472.2 (521.89) | -355.2 (432.04)
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.0393, ANOVA — [p-value comment as in outcome 2, analysis 1]; Treatment as a fixed effect and baseline of the variable predicted as a covariate; least-square means difference = -137.6, 95% CI 2-sided [-268.5 to -6.8]

7. Secondary Outcome: Change From Baseline at 24 Hours in the Tonsillo-Pharyngitis Assessment (TPA) Scores in Participants With Baseline TPA Scores >=8
Description: Tonsillo-Pharyngitis Assessment, or TPA, is an index of seven clinical features of the pain-producing condition itself, pharyngeal inflammation. The clinical features concern temperature, oropharyngeal color, size of tonsils, number of enanthems, largest size of cervical lymph node, number of lymph nodes, and maximum tenderness of lymph nodes. Each variable was rated on a scale of 0-3, with 0 representing the normal value, and 3 representing severe inflammation. The seven values are added together to create the TPA, ranging from 0-21.
  Negative change values represent improvement of symptoms.
Time Frame: Baseline (pre-dose), 24 hours post-dose
Population: Intent to treat population of participants whose baseline TPA was >=8 and had an assessment at hour 24.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 79 | 83
units on a scale | -1.2 (2.61) | -2.0 (2.71)
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.0459, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]

8. Secondary Outcome: Practitioner's Assessment of Pharyngeal Inflammation (P.A.I.N.) Scores at 24 Hours After Initial Dose
Description: P.A.I.N is a four step scale in which physicians rate the severity of pharyngeal inflammation: No inflammation, mild, moderate and severe inflammation.
Time Frame: 24 hours post-dose
Population: Intent to treat population. Three participants withdrew before the 24 hour assessment.
Measure: Number; unit: participants
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 101 | 100
participants
  No inflammation | 0 | 1
  Mild inflammation | 48 | 42
  Moderate inflammation | 42 | 50
  Severe inflammation | 11 | 7
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.8383, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]

9. Secondary Outcome: Investigators' Clinical Assessment (CLIN) Of Study Medication as a Treatment for Sore Throat at 24 Hours After Initial Dose
Description: Investigators assessed the effectiveness of study medication on the patient's sore throat at 24 hours following initial dose by answering the following question: "Considering the patient's response to the study medicine over the past 24 hours, how do you rate the study medicine as a treatment for sore throat?" Responses were poor, fair, good, very good or excellent.
Time Frame: 24 hours
Population: Intent to treat population. Three participants withdrew before the 24 hour assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 101 | 100
percentage of participants
  Poor | 15.8 | 38.0
  Fair | 34.7 | 28.0
  Good | 19.8 | 18.0
  Very Good | 13.9 | 13.0
  Excellent | 15.8 | 3.0
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.0005, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]

10. Secondary Outcome: Participant Satisfaction Scores 24 Hours After Initial Dose
Description: After 24 hours of treatment, participants rated their satisfaction with the treatment on a 7-step scale from extremely dissatisfied to extremely satisfied.
Time Frame: 24 hours
Population: Intent to treat population. Three participants withdrew before the 24 hour assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 101 | 100
percentage of participants
  Extremely dissatisfied | 5.0 | 10.0
  Very dissatisfied | 6.9 | 20.0
  Dissatisfied | 11.9 | 14.0
  Somewhat satisfied | 29.7 | 28.0
  Satisfied | 20.8 | 17.0
  Very satisfied | 23.8 | 9.0
  Extremely satisfied | 2.0 | 2.0
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.0005, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]

11. Secondary Outcome: Investigators' Clinical Assessment (CLIN) Of Study Medication as a Treatment for Sore Throat at the End of the Study (Day 7)
Description: Investigators assessed the effectiveness of study medication on the patient's sore throat at the end of the study by answering the following question: "Considering the patient's response to the study medicine over the past 7 days, how do you rate the study medicine as a treatment for sore throat?" Responses were poor, fair, good, very good or excellent.
Time Frame: Day 7
Population: Intent to treat population of participants who had an end of study assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 93 | 95
percentage of participants
  Poor | 11.8 | 31.6
  Fair | 28.0 | 34.7
  Good | 30.1 | 14.7
  Very Good | 17.2 | 14.7
  Excellent | 12.9 | 4.2
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.0002, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]

12. Secondary Outcome: Time Weighted Sum of Pain Intensity Differences (SPID) in Sore Throat Pain Intensity Scale Over 24 Hours Post-baseline (STPIS SPID24) For Participants With Baseline Practitioner's Assessment of Pharyngeal Inflammation (PAIN) of Moderate or Severe
Description: STPIS measures sore throat pain intensity on a 100-mm visual analog scale completed by participants. A mark at 0-mm indicates no pain upon swallowing and 100-mm indicates severe pain. For the subgroup of patients with moderate/severe pharyngeal inflammation at baseline, SPID24 was calculated as the sum of the time weighted pain intensity differences from baseline until 24 hours. Taking inclusion criteria into account, the full range was -116196 (no pain at any post-dose time (0) - average baseline) to 27804 (maximum possible pain (100) - average baseline).
  Participants with their last recorded time point <21 hours were considered Not Evaluable. If a participant used rescue medication (acetaminophen 650mg was allowed as needed), all post-rescue STPIS values in the 24-hour interval were assigned the baseline value for STPIS. Missing scores of STPIS with non-missing STPIS scores at earlier and later assessments were imputed using linear interpolation.
Time Frame: as for outcome 1
Population: Intent to treat population of participants who took the first full dose of medication and had moderate or severe pharyngeal inflammation at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 68 | 67
units on a scale | -451.4 (491.05) | -283.4 (378.06)
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.0435, ANOVA — [p-value comment as in outcome 2, analysis 1]; least-square means difference = -156.3, 95% CI 2-sided [-307.9 to -4.6]

13. Secondary Outcome: Sore Throat Relief Rating Scale (STRRS) At 2 Hours After Initial Dose
Description: Participants used a 6-category relief scale (no relief to complete relief) to grade the relief of his/her throat pain.
  The patient was instructed to swallow and:
  "Considering how your throat felt before you took the study medicine, circle the phrase that best describes the relief of your sore throat now."
Time Frame: 2 hours
Population: Intent to treat population of participants who had a 2 hour assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 102 | 102
percentage of participants
  No relief | 18.6 | 45.1
  Slight relief | 23.5 | 24.5
  Mild relief | 23.5 | 11.8
  Moderate relief | 20.6 | 13.7
  Considerable relief | 13.7 | 4.9
  Complete relief | 0 | 0
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p < .0001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 2, analysis 1]

14. Secondary Outcome: Time Weighted Sum of Pain Intensity Differences (SPID) in Sore Throat Pain Intensity Scale (STPIS) at Each Post-Dose Time Point Until the Time Point at Which Comparison of the Arms Yielded a P-value <=0.05
Description: Data reported in summary form in Primary Outcome #1 are reported here at each post-dose timepoint until the comparison resulted in a P-value <=0.05 between the two treatment arms.
  STPIS was used to measure sore throat pain intensity using a 100-mm visual analog scale completed by participants that measures "pain on swallowing" (odynophagia). A mark at 0-mm indicates no pain and 100-mm indicates severe pain. The full range of the scale varies by timepoint due to the time weighting sum of SPID. The full scale at 40 minutes post dose was -3188 (complete pain relief within 2 minutes of dosing that lasts 40 minutes) to 812 (maximum pain within 2 minutes lasting 40 minutes) using the mean baseline STPIS.
  If a participant used rescue medication (acetaminophen 650mg was allowed as needed), all post-rescue STPIS values in the 24-hour interval were assigned the baseline value for STPIS. Missing scores of STPIS with non-missing STPIS scores at earlier and later assessments (rec
Time Frame: baseline (pre-dose), up to 23 hours post-dose (every 2 minutes for one hour; every 10 minutes until hour 2; every 30 minutes until hour 6; and every hour the participant was awake between hours 7-23)
Population: Intent to treat population of participants who took the first full dose of medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 102 | 102
units on a scale
  Minutes post dose: 2 | -0.1 (0.26) | -0.2 (0.33)
  Minutes post dose: 4 | -0.3 (0.62) | -0.4 (0.69)
  Minutes post dose: 6 | -0.6 (1.05) | -0.8 (1.14)
  Minutes post dose: 8 | -0.9 (1.56) | -1.2 (1.60)
  Minutes post dose: 10 | -1.4 (2.10) | -1.6 (2.11)
  Minutes post dose: 12 | -1.9 (2.68) | -2.1 (2.59)
  Minutes post dose: 14 | -2.4 (3.30) | -2.5 (3.08)
  Minutes post dose: 16 | -3.0 (3.94) | -2.9 (3.56)
  Minutes post dose: 18 | -3.5 (4.56) | -3.3 (4.01)
  Minutes post dose: 20 | -4.1 (5.19) | -3.7 (4.47)
  Minutes post dose: 22 | -4.7 (5.83) | -4.1 (4.95)
  Minutes post dose: 24 | -5.2 (6.46) | -4.5 (5.43)
  Minutes post dose: 26 | -5.9 (7.12) | -4.9 (5.69)
  Minutes post dose: 28 | -6.5 (7.76) | -5.3 (6.37)
  Minutes post dose: 30 | -7.2 (8.41) | -5.8 (6.87)
  Minutes post dose: 32 | -7.9 (9.09) | -6.2 (7.36)
  Minutes post dose: 34 | -8.6 (9.77) | -6.6 (7.87)
  Minutes post dose: 36 | -9.3 (10.45) | -7.1 (8.37)
  Minutes post dose: 38 | -10.1 (11.14) | -7.5 (8.87)
  Minutes post dose: 40 | -10.8 (11.80) | -7.9 (9.38)
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Minutes post dose: 2; Test type: Superiority or Other; p = 0.1448, ANOVA; Baseline STPIS fitted as a covariate; least-square means difference = 0.1, 95% CI 2-sided [-0.0 to 0.1]
Statistical Analysis 2: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Minutes post dose: 4; Test type: Superiority or Other; p = 0.1538, ANOVA; Baseline STPIS fitted as a covariate; least-square means difference = 0.1, 95% CI 2-sided [-0.0 to 0.3]
Statistical Analysis 3: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Minutes post dose: 6; Test type: Superiority or Other; p = 0.1407, ANOVA; Baseline STPIS fitted as a covariate; least-square means difference = 0.2, 95% CI 2-sided [-0.1 to 0.5]
Statistical Analysis 4: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Minutes post dose: 8; Test type: Superiority or Other; p = 0.2906, ANOVA; Baseline STPIS fitted as a covariate; least-square means difference = 0.2, 95% CI 2-sided [-0.2 to 0.7]
Statistical Analysis 5: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Minutes post dose: 10; Test type: Superiority or Other; p = 0.4758, ANOVA; Baseline STPIS fitted as a covariate; least-square means difference = 0.2, 95% CI 2-sided [-0.4 to 0.8]
Statistical Analysis 6: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Minutes post dose: 12; Test type: Superiority or Other; p = 0.6975, ANOVA; Baseline STPIS fitted as a covariate; least-square means difference = 0.1, 95% CI 2-sided [-0.6 to 0.9]
Statistical Analysis 7: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Minutes post dose: 14; Test type: Superiority or Other; p = 0.9370, ANOVA; Baseline STPIS fitted as a covariate; least-square means difference = 0.0, 95% CI 2-sided [-0.8 to 0.9]
Statistical Analysis 8: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Minutes post dose: 16; Test type: Superiority or Other; p = 0.8493, ANOVA; Baseline STPIS fitted as a covariate; least-square means difference = -0.1, 95% CI 2-sided [-1.1 to 0.9]
Statistical Analysis 9: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Minutes post dose: 18; Test type: Superiority or Other; p = 0.6732, ANOVA; Baseline STPIS fitted as a covariate; least-square means difference = -0.3, 95% CI 2-sided [-1.4 to 0.9]
Statistical Analysis 10: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Minutes post dose: 20; Test type: Superiority or Other; p = 0.5414, ANOVA; Baseline STPIS fitted as a covariate; least-square means difference = -0.4, 95% CI 2-sided [-1.8 to 0.9]
Statistical Analysis 11: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Minutes post dose: 22; Test type: Superiority or Other; p = 0.4313, ANOVA; Baseline STPIS fitted as a covariate; least-square means difference = -0.6, 95% CI 2-sided [-2.1 to 0.9]
Statistical Analysis 12: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Minutes post dose: 24; Test type: Superiority or Other; p = 0.3501, ANOVA; Baseline STPIS fitted as a covariate; least-square means difference = -0.8, 95% CI 2-sided [-2.4 to 0.9]
Statistical Analysis 13: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Minutes post dose: 26; Test type: Superiority or Other; p = 0.2679, ANOVA; Baseline STPIS fitted as a covariate; least-square means difference = -1.0, 95% CI 2-sided [-2.8 to 0.8]
Statistical Analysis 14: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Minutes post dose: 28; Test type: Superiority or Other; p = 0.2137, ANOVA; Baseline STPIS fitted as a covariate; least-square means difference = -1.2, 95% CI 2-sided [-3.2 to 0.7]
Statistical Analysis 15: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Minutes post dose: 30; Test type: Superiority or Other; p = 0.1715, ANOVA; Baseline STPIS fitted as a covariate; least-square means difference = -1.5, 95% CI 2-sided [-3.6 to 0.6]
Statistical Analysis 16: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Minutes post dose: 32; Test type: Superiority or Other; p = 0.1340, ANOVA; Baseline STPIS fitted as a covariate; least-square means difference = -1.8, 95% CI 2-sided [-4.1 to 0.5]
Statistical Analysis 17: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Minutes post dose: 34; Test type: Superiority or Other; p = 0.1030, ANOVA; Baseline STPIS fitted as a covariate; least-square means difference = -2.0, 95% CI 2-sided [-4.5 to 0.4]
Statistical Analysis 18: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Minutes post dose: 36; Test type: Superiority or Other; p = 0.0788, ANOVA; Baseline STPIS fitted as a covariate; least-square means difference = -2.4, 95% CI 2-sided [-5.0 to 0.3]
Statistical Analysis 19: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Minutes post dose: 38; Test type: Superiority or Other; p = 0.0620, ANOVA; Baseline STPIS fitted as a covariate; least-square means difference = -2.7, 95% CI 2-sided [-5.5 to 0.1]
Statistical Analysis 20: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Minutes post dose: 40; Test type: Superiority or Other; p = 0.0476, ANOVA; Baseline STPIS fitted as a covariate; least-square means difference = -3.0, 95% CI 2-sided [-6.0 to -0.0]

15. Secondary Outcome: Kaplan-Meier Estimates for Sore Throat Pain Intensity Scale (STPIS) Time to Definite Improvement
Description: As part of a protocol amendment, some participants defined a definite improvement level (DIL) relative to their actual pretreatment STPIS on the 100-mm visual analog scale. This was done after completing the 7 day trial.
  An alternative definition of STPIS time to onset of relief was the time from initial dose to the time the participant reaching DIL for at least 30 minutes. Data were censored if DIL was not achieved by 120 minutes following initial dose. Definite improvement must also occur prior to re-dosing or using rescue medication.
Time Frame: 2 hours
Population: Intent to treat population of participants who completed the Definite Improvement Level (DIL) following study completion.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 58 | 61
minutes | NA [NA to NA] — Too few participants reached DIL within 2 hours | NA [NA to NA] — Too few participants reached DIL within 2 hours
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.0273, Log Rank

16. Secondary Outcome: Kaplan-Meier Estimates for Sore Throat Pain Intensity Scale (STPIS) Time to Definite Improvement Duration of Relief Using Participant-Defined Definite Improvement Levels (DIL)
Description: As part of a protocol amendment, some participants defined a definite improvement level (DIL) relative to their actual pretreatment STPIS on the 100-mm visual analog scale. This was done after completing the 7 day trial.
  The time of first achieving DIL for 30 minutes within 6 hours (or until rescue or re-dosing) post-dosing will be determined. And the time falling below DIL within 6 hours will be determined. Duration is then defined as the time from first DIL until falling below DIL. Duration was set to zero if the STPIS score does not reach the DIL for at least 30 minutes for STPIS during the 6 hours.
Time Frame: 6 hours
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 58 | 61
minutes | 75.2 (102.41) | 29.4 (65.06)
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.0098, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Initial dose up to Day 7
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/102
Other Adverse Events (participants affected / at risk) | 36/102 | 33/102
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flurbiprofen 8.75 mg Lozenge (N=102) | Placebo Lozenge (N=102)
Tinnitis (Ear and labyrinth disorders) | 1 | 0
Conjunctivitis (Ear and labyrinth disorders) | 1 | 1
Ocular hyperaemia (Ear and labyrinth disorders) | 1 | 0
Abnormal sensation in eye (Ear and labyrinth disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 3 | 2
Oral pain (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 5
Stomatitis (Gastrointestinal disorders) | 2 | 1
Chelilitis (Gastrointestinal disorders) | 1 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 0
Oral discomfort (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Gingival swelling (Gastrointestinal disorders) | 0 | 1
Glossitis (Gastrointestinal disorders) | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 1
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Pain (General disorders) | 0 | 3
Pyrexia (General disorders) | 0 | 2
Tonsillitis (Infections and infestations) | 4 | 3
Otitis media (Infections and infestations) | 3 | 0
Bronchitis (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1
Bite (Injury, poisoning and procedural complications) | 1 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 4 | 0
Headache (Nervous system disorders) | 3 | 6
Paraesthesia oral (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less